CLINICAL TRIAL: NCT02456857
Title: Women's Triple-Negative First-Line Study: A Phase II Trial of Liposomal Doxorubicin, Bevacizumab and Everolimus (DAE) in Patients With Localized Triple-Negative Breast Cancer (TNBC) With Tumors Predicted Insensitive to Standard Neoadjuvant Chemotherapy
Brief Title: Liposomal Doxorubicin, Bevacizumab, and Everolimus in Patients With Locally Advanced TNBC With Tumors Predicted Insensitive to Standard Chemotherapy; A Moonshot Initiative
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2015-0087; NCI-2015-01556 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2015-0087 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2015-05-27; First posted 2015-05-29 (Estimated); Results first posted 2024-02-13 (Actual); Last update posted 2024-02-13 (Actual); Status verified 2024-01

CONDITIONS: Invasive Breast Carcinoma; Triple-Negative Breast Carcinoma
MeSH Terms: conditions — Triple Negative Breast Neoplasms | interventions — Bevacizumab; Immunoglobulin G; Disulfides; Everolimus; liposomal doxorubicin; Doxorubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (DAE) (Experimental): Patients receive pegylated liposomal doxorubicin hydrochloride IV over about 3 hours on day 1, bevacizumab IV over 90 minutes on day 1, and everolimus PO QD on days 1-21. Treatment repeats every 21 days for up to 4 cycles in the absence of disease progression or unacceptable toxicity. Patients will not receive bevacizumab during cycle 4 of therapy. Patients then undergo surgery.
  Interventions: Biological: Bevacizumab; Drug: Everolimus; Other: Laboratory Biomarker Analysis; Drug: Pegylated Liposomal Doxorubicin Hydrochloride

INTERVENTIONS:
Biological: Bevacizumab — Given IV
  Other Names: Anti-VEGF; Anti-VEGF Humanized Monoclonal Antibody; Anti-VEGF rhuMAb; Avastin; Bevacizumab awwb; Bevacizumab Biosimilar BEVZ92; Bevacizumab Biosimilar BI 695502; Bevacizumab Biosimilar CBT 124; Bevacizumab Biosimilar CT-P16; Bevacizumab Biosimilar FKB238; Bevacizumab Biosimilar GB-222; Bevacizumab Biosimilar HD204; Bevacizumab Biosimilar HLX04; Bevacizumab Biosimilar IBI305; Bevacizumab Biosimilar LY01008; Bevacizumab Biosimilar MIL60; Bevacizumab Biosimilar Mvasi; Bevacizumab Biosimilar QL 1101; Bevacizumab Biosimilar RPH-001; Bevacizumab Biosimilar SCT501; Bevacizumab Biosimilar Zirabev; Bevacizumab-awwb; Bevacizumab-bvzr; BP102; BP102 Biosimilar; HD204; Immunoglobulin G1 (Human-Mouse Monoclonal rhuMab-VEGF Gamma-Chain Anti-Human Vascular Endothelial Growth Factor), Disulfide With Human-Mouse Monoclonal rhuMab-VEGF Light Chain, Dimer; Mvasi; Recombinant Humanized Anti-VEGF Monoclonal Antibody; rhuMab-VEGF; SCT501; Zirabev
Drug: Everolimus — Given PO
  Other Names: 42-O-(2-Hydroxy)ethyl Rapamycin; Afinitor; Certican; RAD 001; RAD001; Votubia; Zortress
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Pegylated Liposomal Doxorubicin Hydrochloride — Given IV
  Other Names: ATI-0918; Caelyx; Dox-SL; Doxil; Doxilen; Doxorubicin HCl Liposomal; Doxorubicin HCl Liposome; Doxorubicin Hydrochloride Liposome; Duomeisu; Evacet; LipoDox; Lipodox 50; Liposomal Adriamycin; Liposomal Doxorubicin Hydrochloride; Liposomal-Encapsulated Doxorubicin; Pegylated Doxorubicin HCl Liposome; S-Liposomal Doxorubicin; Stealth Liposomal Doxorubicin; TLC D-99

SUMMARY:
This phase II trial studies how well pegylated liposomal doxorubicin, bevacizumab, and everolimus work in treating patients with triple-negative breast cancer with tumors predicted insensitive to standard chemotherapy. Drugs used in chemotherapy, such as pegylated liposomal doxorubicin, work in different ways to stop the growth of tumor cells by stopping them from dividing. Bevacizumab may stop or slow breast cancer by blocking the growth of new blood vessels necessary for tumor growth. Everolimus may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Giving pegylated liposomal doxorubicin together with bevacizumab and everolimus may kill more tumor cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Determine excellent clinical response rates (pathologic complete response [pCR]/residual cancer burden [RCB]-0 or minimal residual disease [RCB-I]) in patients with anthracycline-based chemotherapy insensitive, localized triple-negative breast cancer (TNBC) who receive 4 cycles of pegylated liposomal doxorubicin hydrochloride, bevacizumab, and everolimus (DAE) following anthracycline-based chemotherapy in the neoadjuvant setting.

SECONDARY OBJECTIVES:

I. Determine response rate after 4 cycles of DAE using radiographic imaging. II. Determine toxicity associated 4 cycles of DAE in the neoadjuvant setting. III. Pathologic response rates to 4 cycles of DAE in mesenchymal tumors versus (vs.) non-mesenchymal tumors.

V. Compare pathologic response rates in mesenchymal tumors to 4 cycles of DAE vs. 12 weeks of weekly paclitaxel (using data collected from standard of care treatment).

EXPLORATORY OBJECTIVES:

I. Determine the correlation between vimentin expression by immunohistochemistry (IHC) and the presence of mesenchymal gene signatures at the time of initial tumor biopsy prior to neoadjuvant chemotherapy (NACT).

II. Determine the correlation between mutations in PIK3CA, PTEN or NF2 or PTEN loss by IHC and the presence of mesenchymal gene signatures at the time of initial tumor biopsy prior to NACT.

III. Determine rates of pCR in patients with mesenchymal tumors identified by gene signatures and compare to pCR rates in non-mesenchymal tumors.

IV. Correlate pathologic response with degree of vimentin expression as measured by IHC.

V. Determine rates of pCR in patients whose tumors contain mutations in PIK3CA, PTEN or NF2 or PTEN loss by IHC and compare to pCR rates in patients whose tumors lacks mutations in these genes.

OUTLINE:

Patients receive pegylated liposomal doxorubicin hydrochloride intravenously (IV) over about 3 hours on day 1, bevacizumab IV over 90 minutes on day 1, and everolimus orally (PO) once daily (QD) on days 1-21. Treatment repeats every 21 days for up to 4 cycles in the absence of disease progression or unacceptable toxicity. Patients will not receive bevacizumab during cycle 4 of therapy. Patients then undergo surgery.

After completion of study treatment, patients are followed up within 30 days of surgery.

ELIGIBILITY:
Inclusion Criteria:

* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Confirmed invasive triple-negative breast cancer defined as estrogen receptor (ER) < 10%; progesterone receptor (PR) < 10% by immunohistochemistry (IHC) and human epidermal growth factor receptor 2 (HER2) 0-1+ (by IHC), or 2+ (fluorescence in situ hybridization [FISH] < 2, gene copy number < 4)
* Primary tumor sample collected before NACT started and
* Undergone molecular testing for integral biomarkers including immunohistochemical staining; the tumor must have evidence of mesenchymal differentiation defined as metaplastic breast cancer, or vimentin >= 50% by IHC
* Received at least one dose of an anthracycline-based NACT; patients are eligible if therapy was discontinued due to disease progression or therapy intolerance
* At least 1.0 cm of measurable residual disease after neoadjuvant anthracycline-based chemotherapy
* Baseline multi-gated acquisition (MUGA) scan or echocardiogram showing left ventricular ejection fraction (LVEF) >= 50% at least 6 weeks prior to initiation of NACT
* Absolute neutrophil count (ANC) >= 1.5 x 10^9/L
* Platelets >= 100 x 10^9/L
* Hemoglobin (Hb) > 9 g/dL
* Total serum bilirubin =< 2.0 mg/dL
* Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) =< 2.5 x upper limit of normal (ULN) (=< 5 x ULN in patients with liver metastases)
* International normalized ratio (INR) =< 2
* Serum creatinine =< 1.5 x ULN
* Fasting serum cholesterol =< 300 mg/dL OR =< 7.75 mmol/L, AND fasting triglycerides =< 2.5 x ULN; NOTE: In case one or both of these thresholds are exceeded, the patient can only be included after initiation of appropriate lipid lowering medication
* Signed informed consent obtained prior to any screening procedures

Exclusion Criteria:

* Pregnant or lactating woman
* Presence of metastatic disease
* Prior therapy with bevacizumab, liposomal doxorubicin, or everolimus
* Prior radiation therapy of the primary breast carcinoma or axillary lymph nodes
* Patients who have a history of another primary malignancy, with the exceptions of: non-melanoma skin cancer, and carcinoma in situ of the cervix, uterus, or breast from which the patient has been disease free for =< 3 years
* Prior cumulative dose of doxorubicin of greater than 360 mg/m^2 or epirubicin of greater than 640 mg/m^2
* Any serious medical illness, other than treated by this study, which would limit survival to less than 1 month or psychiatric illness which would limit informed consent
* Patients with history of serious cardiac events defined as: New York Heart Association class 3 or 4 heart failure, history of myocardial infarction, unstable angina, or cardiovascular accident (CVA) within 6 months of protocol registration; history of PR prolongation or atrioventricular (AV) block
* Known intolerance or hypersensitivity to rapamycin analogs (e.g. sirolimus, temsirolimus)
* Known impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of oral everolimus
* Uncontrolled diabetes mellitus as defined by hemoglobin A1c (HbA1c) > 8% despite adequate therapy; patients with a known history of impaired fasting glucose or diabetes mellitus (DM) may be included, however blood glucose and antidiabetic treatment must be monitored closely throughout the trial and adjusted as necessary
* Patients who have any severe and/or uncontrolled medical conditions such as: a. serious uncontrolled cardiac arrhythmia, or any other clinically significant cardiac disease b. active (acute or chronic) or uncontrolled severe infection, liver disease such as cirrhosis, decompensated liver disease, and active and chronic hepatitis (i.e. quantifiable hepatitis B virus [HBV]-deoxyribonucleic acid [DNA] and/or positive surface antigen of the hepatitis B virus [HBsAg], quantifiable hepatitis C virus [HCV]-ribonucleic acid [RNA]), c. known severely impaired lung function (spirometry and Diffusing capacity of the lungs for carbon monoxide [DLCO] 50% or less of normal and oxygen (O2) saturation 88% or less at rest on room air), d. active, bleeding diathesis; e. Moderate or severe hepatic impairment (Child-Pugh B or C)
* Chronic treatment with corticosteroids or other immunosuppressive agents; topical or inhaled corticosteroids are allowed
* Known history of human immunodeficiency virus (HIV) seropositivity
* Patients who have received live attenuated vaccines within 1 week of start of everolimus and during the study; patient should also avoid close contact with others who have received live attenuated vaccines; examples of live attenuated vaccines include intranasal influenza, measles, mumps, rubella, oral polio, bacillus Calmette-Guerin (BCG), yellow fever, varicella and TY21a typhoid vaccines
* Patients with a history of non-compliance to medical regimens or who are considered potentially unreliable or will not be able to complete the entire study
* Patients who are currently part of or have participated in any clinical investigation with an investigational drug within 1 month prior to dosing
* Women of child-bearing potential (WOCBP), defined as all women physiologically capable of becoming pregnant, must use highly effective methods of contraception during the study and 8 weeks after; highly effective contraception methods include combination of any two of the following:

  * Placement of an intrauterine device (IUD) or intrauterine system (IUS);
  * Barrier methods of contraception: condom or occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/vaginal suppository;
  * Total abstinence or;
  * Male/female sterilization.
  * Note: Women are considered post-menopausal and not of child-bearing potential if they have had 12 months of natural (spontaneous) amenorrhea with an appropriate clinical profile (e.g. age appropriate, history of vasomotor symptoms) or have had surgical bilateral oophorectomy (with or without hysterectomy) or tubal ligation at least six weeks prior to treatment; in the case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment is she considered not of child-bearing potential
* Male patients whose sexual partner(s) are WOCBP who are not willing to use adequate contraception, during the study and for 8 weeks after the end of treatment

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2016-01-12 (Actual); Primary Completion 2023-05-24 (Actual); Study Completion 2023-05-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinton Yam, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Abuhadra N, Sun R, Bassett RL Jr, Huo L, Chang JT, Teshome M, Clayborn AR, White JB, Ravenberg EE, Adrada BE, Candelaria RP, Yang W, Ding Q, Symmans WF, Arun B, Damodaran S, Koenig KB, Layman RM, Lim B, Litton JK, Thompson A, Ueno NT, Piwnica-Worms H, Hortobagyi GN, Valero V, Tripathy D, Rauch GM, Moulder S, Yam C. Targeting chemotherapy resistance in mesenchymal triple-negative breast cancer: a phase II trial of neoadjuvant angiogenic and mTOR inhibition with chemotherapy. Invest New Drugs. 2023 Jun;41(3):391-401. doi: 10.1007/s10637-023-01357-4. Epub 2023 Apr 12. PMID 37043123
- See also: M D Anderson Cancer Center — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment took place in the Breast Medical Oncology clinics of MD Anderson Cancer Center locations during January of 2016 through January of 2020
Groups:
- Liposomal Doxorubicin + Bevacizumab + Everolimus: Liposomal doxorubicin IV 30mg/m2 + Bevacizumab IV (10-15mg/kg) + Everolimus PO 7.5mg
Period: Overall Study
Arm/Group | Liposomal Doxorubicin + Bevacizumab + Everolimus
Started | 17
Completed | 13
Not Completed | 4
Not completed — Disease Progression | 4

BASELINE CHARACTERISTICS:
Arm/Group | Liposomal Doxorubicin + Bevacizumab + Everolimus
Number analyzed (Participants) | 17
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 14
  >=65 years | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 15
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 10
  More than one race | 2
  Unknown or Not Reported | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 17

OUTCOME MEASURES:

1. Primary Outcome: RCB Status
Description: Residual Disease at the time of surgery
Time Frame: up to 3 years
Measure: Number; unit: participants
Arm/Group | Liposomal Doxorubicin + Bevacizumab + Everolimus
Number analyzed (Participants) | 17
participants
  pcR (Best) | 0
  RCB-I | 1
  RCB-II | 13
  RCB-III (Worst) | 3

ADVERSE EVENTS:
Time Frame: 3 years
Arm/Group | Liposomal Doxorubicin + Bevacizumab + Everolimus
All-Cause Mortality (participants affected / at risk) | 0/17
Serious Adverse Events (participants affected / at risk) | 5/17
Other Adverse Events (participants affected / at risk) | 15/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Liposomal Doxorubicin + Bevacizumab + Everolimus (N=17)
Hypertension (Cardiac disorders) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1)
Skin infection (Infections and infestations) | 1 (1)
Pain (General disorders) | 1 (2)
Allergic reaction (General disorders) | 1 (1)
Fever (General disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Liposomal Doxorubicin + Bevacizumab + Everolimus (N=17)
Neutrophil Count Decreased (Investigations) | 4
Anemia (Blood and lymphatic system disorders) | 3
Oral mucositis (Gastrointestinal disorders) | 5
Rash (Skin and subcutaneous tissue disorders) | 2
Headache (Nervous system disorders) | 2
Anorexia (Metabolism and nutrition disorders) | 1
High cholesterol (Infections and infestations) | 1
Creatinine increased (Metabolism and nutrition disorders) | 1
Anxiety (General disorders) | 1
Fatigue (General disorders) | 1
Hypergylcemia (Metabolism and nutrition disorders) | 1
Hypertriglyceridemia (Metabolism and nutrition disorders) | 1
Insomnia (General disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Nail Loss (Skin and subcutaneous tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-02-01): https://cdn.clinicaltrials.gov/large-docs/57/NCT02456857/Prot_SAP_000.pdf